CLINICAL TRIAL: NCT03022175
Title: A Two-part, Double-blind, Placebo-controlled, Phase I Study of the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of SPR741 in Healthy Volunteers
Brief Title: A First in Human Study of the Safety and Tolerability of Single and Multiple Doses of SPR741 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Collaborators: CPR Pharma Services Pty Ltd, Australia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPR741-101s
Record Dates: First submitted 2016-12-16; First posted 2017-01-16 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Healthy Volunteers
Keywords: Safety; Tolerability; Pharmacokinetics
MeSH Terms: interventions — SPR741; Sodium Chloride; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPR741 (Experimental): SPR741 is a novel chemical entity known as a potentiator that specifically interacts with the outer membrane of Gram-negative bacteria to increase the membrane's permeability. This increase in permeability allows Gram-positive antibiotics to enter and kill the cell.
  SAD cohorts: Subjects will receive single doses of SPR741 over 60 minute IV infusion. Planned doses to be studied are 5, 15, 50, 100, 200, 400, 600 and 800 mg.
  MAD cohorts: Subjects will receive SPR741 over 60 minute IV infusion three times a day (TID). Four dose groups will be studied. Doses will be determined by assessing SAD cohort data.
  Interventions: Drug: SPR741
- Placebo (Placebo Comparator): The placebo used during this study is normal saline (0.9% sodium chloride for injection).
  SAD: Subjects will receive single infusions of placebo (0.9% sodium chloride for injection) over 60 minutes.
  MAD: Subjects will receive TID infusions of placebo over 60 minutes for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPR741 — SAD: Double-blind dosing will occur in cohorts 1 through 8. Six participants will receive single doses of SPR741. The dose escalation steps may be altered following review of the safety data upon completion of each cohort.
  MAD: The Safety Management Group will evaluate the safety and tolerability data obtained for the participants in Cohorts 1-5 to determine the appropriate dose level of intravenous q8h dosing of SPR741 to be utilized in the first cohort (Cohort 9) in the MAD. Dosing will commence on the morning of Day 1. Three doses will be administered per day at approximately 8 hours apart. Daily dosing will continue for a total of 14 consecutive days.
  Arms: SPR741
Drug: Placebo — 0.9% sodium chloride for injection. SAD: Two participants in each cohort will receive matching placebo. MAD: Two participants in each cohort will receive matching placebo.
  Other Names: 0.9% sodium chloride for injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of single and multiple intravenous doses of SPR741 when administered to healthy adult volunteers.

DETAILED DESCRIPTION:
This Phase 1 First in Human study is designed to assess the safety, tolerability and pharmacokinetics of single and multiple intravenous doses of SPR741 when administered to healthy adult volunteers. This is a double-blind, placebo controlled, ascending dose, multi-cohort trial. A total of ninety-six healthy volunteers will be enrolled in 12 cohorts. The study will be conducted in two phases: a single ascending dose (SAD) phase, followed by a multiple ascending dose (MAD) phase. In SAD, participants will receive one dose of SPR741 or placebo. In MAD, participants will receive multiple doses of SPR741 or placebo for 14 consecutive days. In both parts, sequential cohorts will be exposed to increasing doses of SPR741.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males and/or females (of non-child bearing potential), 18 to 55 years of age (inclusive) at the time of screening;
2. BMI ≥ 18.5 and ≤ 29.9 (kg/m2) and weight between 62.5 and 100.0 kg (inclusive) for Cohort 1 only and 55.0 and 100.0 kg (inclusive) for all other cohorts;
3. Medically healthy without clinically significant abnormalities at the screening visit or Day -1, including:

   1. Physical examination, vital signs. Vital signs include temperature, heart rate, respiratory rate, and blood pressure;
   2. Triplicate ECGs without QTcF interval duration greater than 450 msec obtained as an average from the triplicate screening and pre-dose Day 1 ECGs after at least 5 min in a fully supine quiet rest;
   3. Hemoglobin/hematocrit, white blood cell (WBC) count, and platelet count greater than the lower limit of normal range of the reference laboratory;
   4. Creatinine, BUN, ALT and AST equal to or less than the upper limit of normal for the reference laboratory; results of all other clinical chemistry and urine analytes without any clinically significant abnormality.

   Discussion between the PI and the SMR is encouraged regarding any abnormal laboratory value that is outside of the normal range during the pre-dose period.
4. Be non-smokers (including tobacco, e-cigarettes or marijuana) for at least 1 month prior to participation in the study;
5. Willing and able to provide written informed consent;
6. Be willing and able to comply with all study assessments and adhere to the protocol schedule;
7. Have suitable venous access for drug administration and blood sampling;
8. If female, be of non-childbearing potential (e.g. post-menopausal as demonstrated by FSH or surgical sterilization i.e., tubal ligation or hysterectomy). Provision of documentation is not required for female sterilization, verbal confirmation is adequate; • If male, a willingness not to donate sperm and if engaging in sexual intercourse with a female partner who could become pregnant, a willingness to use a condom in addition to having the female partner use a highly effective method of birth control (such as an intrauterine device, diaphragm, oral contraceptives, injectable progesterone, subdermal implants, or a tubal ligation). This criterion applies to males (and/or female partners) who are surgically sterile and must be followed from the time of first study drug administration until 30 days after the final administration of study drug.

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or surgery within the past three months determined by the PI to be clinically relevant;
2. History of known or suspected Clostridium difficile infection;
3. Positive urine drug/alcohol testing at screening or check-in (Day -1);
4. Positive testing for HIV, HBsAg or HCV;
5. History of substance abuse or alcohol abuse (defined as greater than 2 standard drinks on average each and every day, where one standard drink is defined as containing 10 g of alcohol and is equivalent to 1 can or stubby of mid-strength beer, 30 ml nip spirits, or 100 ml wine) within the previous 5 years;
6. Use of any prescription medication or any over-the-counter medication, including herbal products and vitamins within 7 days prior to randomization;
7. Documented hypersensitivity reaction or anaphylaxis to any medication;
8. Donation of blood or plasma within 30 days prior to randomization, or loss of whole blood of more than 500 mL within 30 days prior to randomization, or receipt of a blood transfusion within 1 year of study enrollment;
9. Participation in another investigational clinical trial within 30 days prior to Day 1;
10. Any other condition or prior therapy, which, in the opinion of the PI, would make the volunteer unsuitable for this study, including unable to cooperate fully with the requirements of the study protocol or likely to be non-compliant with any study requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-12; Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Safety measures: adverse events | SAD: 5 to 7 days MAD: 21 to 23 days
  The frequency and type of adverse events
Safety measures: clinical laboratory testing | SAD: Day -1 to day 7; MAD: Day -1 to day 21
  Clinical laboratory testing - change from baseline to end of study visit
Safety measures: pulse rate | SAD: Day -1 to day 7; MAD: Day -1 to day 21
  Change from baseline to end of study visit
Safety measures: EKG | SAD: 5 to 7 days MAD: 21 to 23 days
  Change from baseline to end of study visit
Safety measures: respiratory rate | SAD: Day -1 to day 7; MAD: Day -1 to day 21
  Change from baseline to end of study visit
Safety measures: blood pressure | SAD: Day -1 to day 7; MAD: Day -1 to day 21
  Change from baseline to end of study visit

SECONDARY OUTCOMES:
Individual SPR741 plasma concentration-time curves will be tabulated for each dose cohort. | Day 1 and Day 14
  • Blood draws for PK: pre-dose (within 10 minutes), 30 minutes following the start of infusion, end of infusion and at 90, 150 minutes, 3, 4, 5, 6 and 8 hours following start of infusion (Day 1 (first dose) and Day 14 (last dose)). Five additional blood draws will be obtained at 10, 12, 24, 36 and 48 hours following the start of infusion of the last dose (morning of Day 14).
Geometric means will be calculated for Area Under the Curve (AUC) | Day 1 and Day 14
  Blood draws for PK: pre-dose (within 10 minutes), 30 minutes following the start of infusion, end of infusion and at 90, 150 minutes, 3, 4, 5, 6 and 8 hours following start of infusion (Day 1 (first dose) and Day 14 (last dose)). Five additional blood draws will be obtained at 10, 12, 24, 36 and 48 hours following the start of infusion of the last dose (morning of Day 14).
Geometric means will be calculated for Concentration maximum (Cmax) | Day 1 and Day 14
  Blood draws for PK: pre-dose (within 10 minutes), 30 minutes following the start of infusion, end of infusion and at 90, 150 minutes, 3, 4, 5, 6 and 8 hours following start of infusion (Day 1 (first dose) and Day 14 (last dose)). Five additional blood draws will be obtained at 10, 12, 24, 36 and 48 hours following the start of infusion of the last dose (morning of Day 14).
Geometric means will be calculated for Area Under the Curve (AUC) Urine | Day 1 and Day 14
  • Urine collection for PK: pre-dose Day 1 sample, total collection over 0-4, 4-8 hours following start of infusion of first dose on Day 1; then total collection over 0-4, 4-8, 8-12, 12-24 and 24-48 hours following start of infusion of the last dose (Day 14).
Geometric means will be calculated for Concentration maximum (Cmax) Urine | Day 1 and Day 14
  • Urine collection for PK: pre-dose Day 1 sample, total collection over 0-4, 4-8 hours following start of infusion of first dose on Day 1; then total collection over 0-4, 4-8, 8-12, 12-24 and 24-48 hours following start of infusion of the last dose (Day 14).
Mean SPR741 plasma concentration-time curves will be tabulated for each dose cohort. | Day 1 and Day 14
  • Blood draws for PK: pre-dose (within 10 minutes), 30 minutes following the start of infusion, end of infusion and at 90, 150 minutes, 3, 4, 5, 6 and 8 hours following start of infusion (Day 1 (first dose) and Day 14 (last dose)). Five additional blood draws will be obtained at 10, 12, 24, 36 and 48 hours following the start of infusion of the last dose (morning of Day 14).

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Farinola, MB, BSc, FRACP, Principal Investigator — CMAX - A division of IDT Australia, Limited
Locations (1):
- CMAX - A division of IDT Australia, Limited, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eckburg PB, Lister T, Walpole S, Keutzer T, Utley L, Tomayko J, Kopp E, Farinola N, Coleman S. Safety, Tolerability, Pharmacokinetics, and Drug Interaction Potential of SPR741, an Intravenous Potentiator, after Single and Multiple Ascending Doses and When Combined with beta-Lactam Antibiotics in Healthy Subjects. Antimicrob Agents Chemother. 2019 Aug 23;63(9):e00892-19. doi: 10.1128/AAC.00892-19. Print 2019 Sep. PMID 31262767